CLINICAL TRIAL: NCT04153383
Title: Milrinone on Cardiac Performance in Patients Undergoing Off-pump Coronary Artery Bypass Surgery
Brief Title: Milrinone on Cardiac Performance During Off-pump Coronary Artery Bypass Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Konkuk University Medical Center (Other)
Responsible Party: Principal Investigator, Tae-Yop Kim, MD PhD, Professor of Anesthesiology, Konkuk University Medical Center
Other Study IDs: KUH0000000123
Record Dates: First submitted 2019-11-04; First posted 2019-11-06 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Ischemic Heart Disease
Keywords: Milrinone; diastolic function
MeSH Terms: conditions — Myocardial Ischemia | interventions — Milrinone

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TMAD: Tissue motion annular displacement (TMAD) of tricuspid valve annulus transesophageal echocardiography
  Interventions: Drug: Milrinone Injection

INTERVENTIONS:
Drug: Milrinone Injection — giving IV milrinone: 50 mcg/kg loading dose by IV push over 10 minutes, then 0.375-0.75 mcg/kg/min IV
  Other Names: Milrinone

SUMMARY:
The purpose of this study is to analyze the changes in cardiac performance before and after milrinone administration in order to find out whether milrinone improves LV performance in patients undergoing coronary artery bypass surgery.

ELIGIBILITY:
Inclusion Criteria:

* patient agree and provide written informed consent.
* patient undergoing elective coronary artery bypass graft surgery
* preoperative LV EF>50% (TTE)

Exclusion Criteria:

* preoperative cardiac dysrhythmia
* preoperative IABP
* use of other inotropic agents

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: valvular heart disease
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
TMAD of ticuspid annulus during early relaxation | 15 mini after milrinone administration

SECONDARY OUTCOMES:
global longitudinal strain of the right ventricle | 15 mini after milrinone administration
left ventricular ejection fraction | 15 min after milline administration
global longitudinal strain of the left ventricle | 15 min after milline administration